CLINICAL TRIAL: NCT04730362
Title: Effect of Laryngeal Mask Airway on Image Quality n Pediatric Patients Undergoing Magnetic Resonant Imaging: a Randomized Controlled Trial
Brief Title: Effect of Laryngeal Mask Airway on Image Quality n Pediatric Patients Undergoing Magnetic Resonant Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Abdelfattah Abdelwadod, Mohammed Abdelfattah Abdelwadod, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2007-50111
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: Control group : a Guedel oral airway will be inserted for airway management versus supraglottic group patients in which supraglottic airway laryngeal mask airway (LMA) will be used
Who Masked: Participant, Investigator
Masking Description: Randomization is done using computer generated sequence. Concealment will be achieved by opaque envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 20 patients in which a Guedel oral airway will be inserted for airway management and to conduct inhalational anesthetic through face mask fixed with harness to the head and then connected to anesthesia breathing circuit of MRI compatible anesthesia machine for maintenance of anesthesia of O2 and sevoflurane 2-4% .
  Interventions: Device: guedel airway; Drug: propofol bolus and then anesthesia sevoflurane
- supraglottic group (Active Comparator): 20 patients in which supraglottic airway laryngeal mask airway (LMA) will be used and then connected to anesthesia breathing circuit of MRI compatible anesthesia machine for maintenance of anesthesia of O2 and sevoflurane 2-4% .
  Interventions: Device: supraglottic airway; Drug: propofol bolus and then anesthesia sevoflurane

INTERVENTIONS:
Device: guedel airway — Anesthesia will be conducted by induction with 1-2
  • Mg/kg of an IV propofol bolus and then anesthesia is maintained with an inhalational anesthesia with sevoflurane 2%-4%. The goal is to maintain the patient spontaneous ventilation throughout the procedure. Monitoring of the patients is done by MRI compatible pulse oximetry for heart rate and oxygen saturation which is connected to MRI control room.
  Arms: Control group
Device: supraglottic airway — supraglottic airway
  Arms: supraglottic group
Drug: propofol bolus and then anesthesia sevoflurane — Mg/kg of an IV propofol bolus and then anesthesia is maintained with an inhalational anesthesia with sevoflurane 2%-4%

SUMMARY:
This study compare the effects of Oral airway vs LMA in preventing anesthesia-induced partial airway obstruction, in an attempt to lessen MRI motion artifacts, which would result in improvements in image quality.

DETAILED DESCRIPTION:
Magnetic resonance image (MRI) is a frequently used imaging technique especially in oncological patients, where it is used for diagnosis, following up response to treatment and later for detection of possible recurrence. The main problem encountered with MRI is the long time required for completion of the imaging, during which the patient is required to lie still. Patients who are unable to lie still require sedation or general anesthesia (GA). Almost all pediatric patients are uncooperative, making GA, the standard of care for pediatric MRI.

Several general anesthetic techniques including airway management by endotracheal tube & various supraglottic devices (LMA) have been described. Choice of technique by anesthesiologist is influenced by the patient's age, craniofacial and airway anatomy, procedure duration, & illness acuity.

ELIGIBILITY:
Inclusion Criteria:

* ASA І and II patients
* Age under 18 years .
* The patient will need GA and patient Scheduled for MRI brain.

Exclusion Criteria:

* Glasgow coma scale ≤ 8
* Emergency patient with full stomach.
* Distorted upper airway anatomy making intubation with GA mandatory.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Image quality of each MRI sequence | During general anesthesia of MRI investigation procedure
  Image quality of each MRI sequence is evaluated by using a scoring system with the following scores: score of 1 (non-diagnostic), score of 2 (poor quality but some diagnostic value), score of 3 (average), score of 4 (good), and score of 5 (excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Nataional Cancer Instituite, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided